CLINICAL TRIAL: NCT04021446
Title: A Supervised Clinic-to-Community Exercise Intervention to Improve Cardiometabolic Health in Survivors of Adolescent and Young Adult Cancer: The ACSEND Trial
Brief Title: A Supervised Clinic-to-Community Exercise Intervention to Improve Cardiometabolic Health in Survivors of AYA Cancer
Acronym: ASCEND
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, Assistant Professor of Research, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AYA_ASCEND
Record Dates: First submitted 2019-03-12; First posted 2019-07-16 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cardiometabolic Dysregulation; Young Adult Cancer; Adolescent Cancer; Body Composition
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): Will receive the exercise intervention
  Interventions: Other: Exercise
- Attention Control (No Intervention): Will not receive the exercise intervention

INTERVENTIONS:
Other: Exercise — personalized exercise prescription
  Arms: Exercise

SUMMARY:
The main goal of this clinical trial is to use a novel exercise intervention to improve cardiometabolic and biopsychosocial health outcomes in overweight/obese sedentary survivors of AYA cancers at risk for chronic comorbid conditions. The investigator's hypothesis is that an exercise intervention will improve: cardiometabolic health; body composition; physical fitness and biopsychosocial outcomes when compared to the attention control group.

ELIGIBILITY:
Inclusion Criteria:

* AYA cancer survivors (18-39) Must be 12 months after treatment No metastatic disease

Exclusion Criteria:

* Metastatic disease Pregnancy

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Cardiometabolic health - Insulin Resistance | change from baseline to 4 months, to 8 months to 1 year
  insulin resistance estimated by HOMA from a fasting blood sample
Cardiometabolic health - metabolic syndrome waist circumference | change from baseline to 4 months, to 8 months to 1 year
  markers of metabolic syndrome, waist circumference via measuring tape (cm)
Cardiometabolic health - metabolic syndrome blood pressure | change from baseline to 4 months, to 8 months to 1 year
  markers of metabolic syndrome, blood pressure via Omron cuff (mmHg)

SECONDARY OUTCOMES:
Body Composition | change from baseline to 4 months, to 8 months to 1 year
  fat mass and lean mass via DEXA (reported in lbs)
Cardiorespiratory fitness (Physical Fitness) | change from baseline to 4 months, to 8 months to 1 year
  cardiorespiratory fitness via submaximal VO2 max (reported via ml/kg/min)
Muscular Strength (Physical Fitness) | change from baseline to 4 months, to 8 months to 1 year
  muscle strength through multiple repetition maximum (lbs)